CLINICAL TRIAL: NCT04277663
Title: A Phase 3, Open-label, Multicenter Study, IBI310 in Combination With IBI308 and IBI308 Compared to High-Dose Interferon In Patients With Acral Melanoma That Has Been Removed by Surgery
Brief Title: The Study of IBI310 in Combination With IBI308 Compared to High-Dose Interferon In Patients With Acral Melanoma That Has Been Removed by Surgery
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to the company's development strategy adjustment ，Innovent Bioligics decided not to continue the study after consultation with investigators
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIBI310A301
Record Dates: First submitted 2020-02-18; First posted 2020-02-20 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Acral Melanoma That Has Been Removed by Surgery
MeSH Terms: interventions — sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IBI310 + IBI308 (Experimental): Participants will be treated with IBI310 in combination with IBI308
  Interventions: Drug: IBI310+IBI308
- IBI308 (Experimental): Participants will be treated with IBI308
  Interventions: Drug: IBI308
- high-dose recombinant interferon a-2B (Active Comparator): Participants will be treated with recombinant interferon a-2B
  Interventions: Drug: High-dose recombinant interferon a-2B

INTERVENTIONS:
Drug: IBI310+IBI308 — In this group, subjects will be given IBI310 3mg/kg IV Q3W in combination with IBI308 200mg IV Q3W for 4 cycles, then follow up a maintenance therapy performed with IBI310 3mg/kg IV Q12W in combination with IBI308 200mg IV Q3W until disease progression or loss of clinical benefit.
  Arms: IBI310 + IBI308
Drug: IBI308 — In this group, subjects will be given IBI308 200mg IV Q3W until disease progression or loss of clinical benefit
  Arms: IBI308
Drug: High-dose recombinant interferon a-2B — In this group, subjects will be given 15*10^9 U/m2/d recombinant interferon a-2B intravenously on days 1-5 weekly for 4 weeks.Then 9*10^9 U/m2/d recombinant interferon a-2B intravenously three times weekly for 48 weeks
  Arms: high-dose recombinant interferon a-2B

SUMMARY:
This is a phase III randomized, control, multi-center study of recombinant humanized anti-PD-1 mAb in combination with CTLA4 mAb for injection compared to high-Dose interferon in patients with acral melanoma that has been removed by surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the written informed consent (Informed Consent, ICF), and be able to abide by the visits and related procedures stipulated in the plan.
2. Completely resected stage IIIB-IV acral melanoma (according to the 8th edition of AJCC staging criteria for malignant melanoma of the skin). Complete resection of stage III melanoma includes extended resection of the primary lesion and/or regional lymph node dissection and/or resection of satellite nodules. Complete resection of stage IV melanoma includes resection of primary tumor and complete resection of metastases. Complete resection of melanoma should conform to the principle of R0 resection and be confirmed by the investigator. Requirements for regional lymph node dissection refer to: upper extremity melanoma, at least 10 lymph nodes in the draining lymph node area; lower extremity melanoma, at least 5 lymph nodes in the draining lymph node area. In special cases, such as ① the long diameter of lymph nodes is ≥ 3 cm, it is considered that the number of lymph nodes can not be resected because of lymph node fusion; ② the draining lymph node area that needs to be cleaned only includes the cubital fossa or popliteal fossa, and the number of lymph nodes is difficult to reach 5-10, etc., it needs to be studied The patient confirmed whether the lymph node dissection was in line with R0 resection.
3. Stage IIIB-IV acral melanoma with histologically/cytologically confirmed primary lesions in extremities (hands, feet, subungual nails). For subjects with only metastatic lesions confirmed by histopathology, researchers need to confirm that the primary lesions are in the extremities and exclude other primary sites, and they can discuss with the medical monitors to decide whether to enroll.
4. The first study drug injection can only be carried out when the incision is completely healed after melanoma resection, and the injection time should not exceed 13 weeks after the operation (if the time limit is exceeded due to unforeseen reasons, it can be discussed with the medical supervisor decision to enroll).
5. Within 4 weeks before randomization, R0 complete resection was confirmed by physical examination and imaging examination.

Exclusion Criteria：

1. Mucosal-derived melanoma, ocular uveal melanoma, transitional metastasis and leptomeningeal metastasis.
2. Previously exposed to any anti-CTLA-4, anti-PD-1 or anti-PD-L1/2 antibodies.
3. Previous use of interferon. If interferon therapy was used ≥ 1 year before the first dose of study treatment, and the treatment time was ≤ 30 days or the treatment dose was ≤ 3×106IU/d, they could be enrolled.
4. Hyperthyroidism or hypothyroidism, Note: Hypothyroidism subjects with stable condition after hormone replacement therapy can be enrolled.
5. Participate in another clinical study at the same time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2020-04-17 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Recurrence-free survival rate | up to 5 years after enrollment
  to evaluate the Recurrence free survival (RFS) of the patients with acral melanoma treated by IBI310 in Combination With IBI308 and high-Dose interferon

SECONDARY OUTCOMES:
Overall survival (OS) | up to 5 years after enrollment
  to evaluate the Overall survival (OS) of the patients with acral melanoma treated by IBI310 in Combination With IBI308 and high-Dose interferon

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing cancer hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No